CLINICAL TRIAL: NCT02102555
Title: A Double-blind Randomized, Placebo-controlled Study to Determine the Effectiveness of Pre-operative IV Acetaminophen Administration in Reducing Post-operative Pain, Nausea, and Vomiting in the Outpatient Setting
Brief Title: Acetaminophen vs Placebo in the Pre-operative Setting and Outcomes on Post-operative Pain, Nausea and Vomiting
Acronym: IV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: study closed due to difficulty enrolling subjects - no results
Sponsor: MercyOne Des Moines Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMC2013-25
Record Dates: First submitted 2014-01-31; First posted 2014-04-03 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2019-08

CONDITIONS: Post Operative Pain; Post Operative Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Vomiting | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV acetaminophen (Active Comparator): Patients in the IV acetaminophen arm will receive a one gram dose of IV acetaminophen in the pre-operative area prior to their surgery.
  Interventions: Drug: IV acetaminophen
- Placebo (Placebo Comparator): Patients in the placebo arm will receive normal saline in the pre-operative area.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IV acetaminophen — Single dose of one gram of IV acetaminophen given in pre-operative area
  Other Names: Ofirmev; paracetamol
  Arms: IV acetaminophen
Drug: placebo — placebo (IV normal saline)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a single dose of IV acetaminophen can improve post-operative pain, nausea, and vomiting in the outpatient setting. Patient satisfaction, time to readiness of discharge, and the amount of opiates post operatively will also be measured.

DETAILED DESCRIPTION:
The purpose of this study is to determine if using a one time pre-operative dose of IV acetaminophen has an effect on post-operative nausea, vomiting, and pain. This is a randomized, double-blind, placebo-controlled prospective study on patients from the Katzmann Breast Center undergoing outpatient breast surgery (including excisional biopsy, lumpectomy, sentinel lymph node biopsy, axillary node dissection, or ductal excision).

IV acetaminophen (paracetamol) has been in Europe and other countries. In the U.S. the FDA approved IV acetaminophen (Ofirmev) in November of 2010. Since then, it has been used in many different ways, but most commonly in the first 24 hours post operative recovery period.

There will be two arms included in this study. Patients in Arm One will receive a one gram dose of IV acetaminophen in the pre-operative area. Patients in Arm Two will receive a dose of the placebo (IV normal saline). The medication will be disguised in the same bag as the normal saline, so no one (including the patient) in the pre-operative area will know which arm the patient is in. This prospective, randomized, double blind study will compare post-operative nausea, vomiting, and pain rates in patients from both arms.

The primary endpoint of this study will be to compare post-operative pain in patients receiving a pre-operative dose of IV acetaminophen to patients receiving the normal saline placebo. Secondary endpoints will include post-operative nausea and vomiting, recovery times, and overall satisfaction of pain management throughout their experience (assessed on post operative day one). If this study shows that IV acetaminophen given in the pre-operative setting decreases post-operative nausea, vomiting, and/or pain and/or shortens recovery time, and improves patient satisfaction in regards to their pain management, it could also become a routine medication given to all patients in the pre-operative setting.

ELIGIBILITY:
Inclusion Criteria:

Each of the following must be met:

* Greater than or equal to 18 years of age.
* Female
* Undergoing outpatient breast surgery (unilateral or bilateral surgery)

Exclusion Criteria:

If ANY of the following apply:

* History of an allergy or hypersensitivity to acetaminophen (oral, rectal, or IV)
* Chronic alcoholism
* Severe deficiency of liver and/or kidney
* Any patient unable to sign informed consent
* Pregnancy
* Any patient currently enrolled in another experimental protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-10; Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
postoperative pain | first postoperative day
  postoperative pain as measured by visual analog scale (VAS, range 0-10) measured in recovery room before discharge to outpatient setting

SECONDARY OUTCOMES:
postoperative nausea and vomiting (PONV) | first postoperative day
  patient-rated postoperative nausea and vomiting (PONV) on visual analog scale
time until readiness of discharge | first postoperative day
  time until readiness of discharge: measured from arrival to the recover room to discharge-order-written time (DOW time)
IV analgesic consumption in recovery room | first postoperative day
  intravenous analgesic consumption in recovery room: converted to morphine-equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Lauren D Allan, DO, Principal Investigator — Mercy Medical Center-Des Moines General Surgery Residency
Locations (1):
- Mercy Medical Center-Des Moines, Des Moines, Iowa, United States